CLINICAL TRIAL: NCT00257062
Title: A Multicenter, Double-Blind, Randomized Study to Compare the Safety and Efficacy of Oral Levofloxacin With That of Ciprofloxacin HCl in the Treatment of Uncomplicated Skin and Skin Structure Infections in Adults
Brief Title: A Study of the Safety and Effectiveness of Oral Levofloxacin Compared With Oral Ciprofloxacin in the Treatment of Adults With Uncomplicated Infections of the Skin and the Supportive Layers Beneath the Skin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005479
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Skin Diseases, Infectious
Keywords: Infectious skin diseases; skin diseases; bacterial skin diseases; antibacterial agents; quinolones; levofloxacin
MeSH Terms: conditions — Skin Diseases, Infectious; Skin Diseases; Skin Diseases, Bacterial | interventions — Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of levofloxacin, an antibiotic, compared with another antibiotic, ciprofloxacin, in the treatment of adults with uncomplicated infections of the skin and the supportive layers beneath the skin.

DETAILED DESCRIPTION:
Levofloxacin is an antibacterial agent used for the treatment of many types of infections in adults. This is a randomized, double-blind, parallel group, multicenter study to determine the safety and effectiveness of levofloxacin (500 mg once daily for 7 days) compared with ciprofloxacin (500 mg once every 12 hours for 10 days) in adults with uncomplicated infections of the skin and the supportive layers beneath the skin. The study consists of 3 visits: one visit for screening and enrollment, and 2 visits for assessment of safety and effectiveness (one visit on Days 3 - 5 of the study and one visit [post-therapy] 2 - 7 days after the last dose of the study drug). The total duration of patient participation in the study is approximately 2 weeks. The primary assessments of effectiveness include the clinical response to treatment (categorized at post-therapy as cured, improved, or failed) and the microbiological response at post-therapy (the elimination of the disease-causing bacteria, categorized as eradicated, partially eradication, or persisted, determined by patient and by type of bacteria). Safety evaluations (incidence of adverse events, physical examination, and laboratory tests) are performed throughout the study. The study hypothesis is that treatment with levofloxacin is at least as effective and as well tolerated as treatment with ciprofloxacin in patients with uncomplicated infections of the skin and the supportive layers beneath the skin. One levofloxacin 500 mg tablet by mouth, once daily (and a placebo tablet once daily, 12 hours later) for 7 days, followed by one placebo tablet every 12 hours for 3 days; or one ciprofloxacin 500 mg tablet by mouth once every 12 hours for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of infection of the skin and/or the supportive layers beneath the skin, as indicated by pain at the site of the infection, redness, swelling, drainage, or other relevant clinical signs
* able to provide a sample of tissue from the affected area of the skin
* able to receive oral medications.

Exclusion Criteria:

* Patients with a condition requiring treatment with antibiotics by injection into a vein, a muscle, or beneath the skin
* having a severe infection
* previous allergic or serious adverse reaction to similar antibiotics, or have severe lactose intolerance
* taken antibiotics internally within 48 hours of the start of the study with resulting improvement
* requirement of a second antibiotic taken internally or requirement of an antibiotic applied directly to the site of the infection in addition to the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 1993-01; Study Completion 1994-04 (Actual)

PRIMARY OUTCOMES:
Clinical response rate at post-therapy (defined as cured, improved or failed); microbiological response at post-therapy (rate of elimination of disease-causing bacteria, by patient, and by type of bacteria); incidence of adverse events

SECONDARY OUTCOMES:
Changes in physical examination and laboratory tests after treatment with the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the safety and effectiveness of oral levofloxacin compared with oral ciprofloxacin in the treatment of adults with uncomplicated infections of the skin and the supportive layers beneath the skin — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=652&filename=CR005479_CSR.pdf